CLINICAL TRIAL: NCT03061318
Title: Validation of a Multi-Genetic Test for the Diagnosis of Indeterminate Thyroid Nodules
Acronym: CT-DS
Status: Completed | Type: Observational
Sponsor: Hernán González (Other)
Responsible Party: Sponsor-Investigator, Hernán González, Associate Professor -Head and Neck Surgeon, Pontificia Universidad Catolica de Chile
Organization: Pontificia Universidad Catolica de Chile (Other)
Other Study IDs: 14-463
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Indeterminate Thyroid Cytology
Keywords: Fine Needle Aspiration, Genetic Classifier

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Thyroid Nodule Fine Needle Aspiration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A clinical trial is proposed, to clinically validate the diagnostic performance of a new genetic test developed in Chile. It will determine the nature of thyroid nodules that have been informed as indeterminate by cytology through a fine needle aspiration (FNA).

The Genetic Classifier for Indeterminate Thyroid Nodules is a quantitative gene expression test, that combines the results for a panel of 10 biomarkers (CXCR3, CCR3, CXCl10, CK19, TIMP1, CLDN1, CAR, XB130, HO-1 and CCR7), to generate a single number score. It is indicated on patients with a thyroid nodule informed by cytology as indeterminate (Bethesda III and IV, according to The Bethesda System for Reporting Thyroid Cytopathology). This test would be used by taking a sample with a fine needle aspiration (FNA) and thus, being able to predict, with high accuracy, benign nodules that do not require surgery.

DETAILED DESCRIPTION:
Problem/Necessity: Throughout the world, each year, hundreds of thousands of patients undergo an unnecessary diagnostic surgery of the thyroid. This occurs in patients that have a FNA informed as indeterminate (which correspond to 15-20% of all FNA), due to have a risk of malignancy ranging from 15 to 25%. So, 75% of the indeterminate nodules are unnecessarily operated, which makes it essential to have a diagnostic tool that allows us to identify those patients with benign thyroid nodules and thus, avoid surgery.

Solution: We have developed a test that, through the analysis of the expression of 10 genes by PCR on real time in FNA samples, integrated by an algorithm, rules out the presence of cancer with a Negative Predictive Value (NPV) of 96% and Specificity of 81%.

Benefit/Justification: The high NPV will allow the clinician to recommend observation as an alternative to surgery. The 6% of false negatives is clinically accepted due to, cytology on its own, has 5% of false negatives. On the other hand, the 75% of specificity will allow to avoid surgery on 75% of the benign cases, which makes the test cost-effective.

State of Progress: The test has completed the phase of prototype development and analytical validation. The next stage is the clinical validation and it corresponds to the study proposed on this protocol.

Hypothesis: Our genetic test rules out the presence of cancer with a NPV higher that 94% and Specificity higher than 75% on indeterminate nodule samples.

Proposed study: A multi-centric (9 sites) clinical trial will be developed in Chile, with statistical power to determine the sensitivity and clinical specificity, negative and positive predictive values, likelihood ratios and confidence intervals.

Method: Patients that have a FNA indicated by their treating physician, due to they have an indeterminate nodule that requires to be determined if it is benign or malignant, will be invited to participate on this trial. After the informed consent is signed, a FNA sample will be obtained for cytology and for molecular study. Obtaining the sample for the molecular study will be part of the same procedure. A maximum of 4000 samples must be enrolled. Approximately 300 will fulfill all of the requirements to complete the study, which include: having a confirmed indeterminate cytology, be sent to surgery (gold standard), and have a proper mRNA sample. Throughout the study, the treating physician will not modify his conduct at any time and the decisions will be based on the clinical information that is regularly used.

Timeline/Monitoring: The study recruitment phase is expected to last an approximate of 28 months (24 months of enrollment, and 4 months of follow up as a minimum time to obtain the result for the surgical biopsy). However, this timeline might be extended while waiting for the 300 indeterminate samples to end study. There will be a principal investigator on each site, guided by a hired CRO, will guard the correct execution of the trial.

ELIGIBILITY:
Inclusion Criteria:

Patient ≥ 18 years old, male or female Patent with a thyroid nodule ≥ 8.0 mm of diameter measured by ultrasound. Patient with indication of thyroid fine needle aspiration (FNA). Patient with no record of spontaneous bleeding. Patient in condition to understand and sign the ICF.

Exclusion Criteria:

1. Patient < 18 years old, male or female.
2. Patient with an ultrasound diagnosis of thyroid nodule < 8.0 mm.
3. Patient with record of spontaneous bleeding.
4. Patient with current symptoms of bleeding.
5. Patient in no condition of understanding and signing the ICF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be conducted on a patient population that has, according to their treating physicians, the clinical indication of FNA due to the presence of a thyroid nodule. Enough patients will be enrolled to obtain a maximum of 3600 to 4000 FNA. Patients will not be exposed to additional risks, beyond those that may occur as a result of the procedure of Fine Needle Aspiration. Patients that participate on this study, will be exposed to the (minimum) risks associated to the thyroid tissue sample technique by fine needle aspiration.
Sampling Method: Non-Probability Sample
Enrollment: 3100 (Actual)
Dates: Start 2015-08-08 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Verify the sensitivity, specificity, NPV, PPV. | 30 months
  Sensitivity: True Positives Specificity: True Negatives NPV: Ability to predict Benign PPV: Ability to predict Malignant

CONTACTS AND LOCATIONS:
Overall Officials: Hernán E González, MD, Study Director — Pontificia Universidad Catolica de Chile
Locations (9):
- Chile (9):
  - Centro de Diagnóstico Plaza Italia, Santiago, Santiago Metropolitan
  - Clínica Alemana de Santiago, Santiago, Santiago Metropolitan
  - Clínica San Carlos de Apoquindo, Santiago, Santiago Metropolitan
  - Clínica Santa María, Santiago, Santiago Metropolitan
  - Fundación Arturo López Pérez, Santiago, Santiago Metropolitan
  - Hospital Clínico de la Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan
  - Hospital del Salvador, Santiago, Santiago Metropolitan
  - Hospital San Juan de Dios, Santiago, Santiago Metropolitan
  - Hospital Clínico de la Universidad de Chile, Santiago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sipos JA, Mazzaferri EL. Thyroid cancer epidemiology and prognostic variables. Clin Oncol (R Coll Radiol). 2010 Aug;22(6):395-404. doi: 10.1016/j.clon.2010.05.004. Epub 2010 Jun 3. PMID 20627675
- [Background] Pellegriti G, Frasca F, Regalbuto C, Squatrito S, Vigneri R. Worldwide increasing incidence of thyroid cancer: update on epidemiology and risk factors. J Cancer Epidemiol. 2013;2013:965212. doi: 10.1155/2013/965212. Epub 2013 May 7. PMID 23737785
- [Background] Davies L, Welch HG. Current thyroid cancer trends in the United States. JAMA Otolaryngol Head Neck Surg. 2014 Apr;140(4):317-22. doi: 10.1001/jamaoto.2014.1. PMID 24557566
- [Background] Sosa JA, Hanna JW, Robinson KA, Lanman RB. Increases in thyroid nodule fine-needle aspirations, operations, and diagnoses of thyroid cancer in the United States. Surgery. 2013 Dec;154(6):1420-6; discussion 1426-7. doi: 10.1016/j.surg.2013.07.006. Epub 2013 Oct 2. PMID 24094448
- [Background] Bongiovanni M, Spitale A, Faquin WC, Mazzucchelli L, Baloch ZW. The Bethesda System for Reporting Thyroid Cytopathology: a meta-analysis. Acta Cytol. 2012;56(4):333-9. doi: 10.1159/000339959. Epub 2012 Jul 25. PMID 22846422
- [Background] Wang CC, Friedman L, Kennedy GC, Wang H, Kebebew E, Steward DL, Zeiger MA, Westra WH, Wang Y, Khanafshar E, Fellegara G, Rosai J, Livolsi V, Lanman RB. A large multicenter correlation study of thyroid nodule cytopathology and histopathology. Thyroid. 2011 Mar;21(3):243-51. doi: 10.1089/thy.2010.0243. Epub 2010 Dec 29. PMID 21190442
- [Background] Hodak SP, Rosenthal DS; American Thyroid Association Clinical Affairs Committee. Information for clinicians: commercially available molecular diagnosis testing in the evaluation of thyroid nodule fine-needle aspiration specimens. Thyroid. 2013 Feb;23(2):131-4. doi: 10.1089/thy.2012.0320. Epub 2012 Nov 27. PMID 22984796
- [Background] Nikiforova MN, Wald AI, Roy S, Durso MB, Nikiforov YE. Targeted next-generation sequencing panel (ThyroSeq) for detection of mutations in thyroid cancer. J Clin Endocrinol Metab. 2013 Nov;98(11):E1852-60. doi: 10.1210/jc.2013-2292. Epub 2013 Aug 26. PMID 23979959
- [Background] Nikiforov YE, Ohori NP, Hodak SP, Carty SE, LeBeau SO, Ferris RL, Yip L, Seethala RR, Tublin ME, Stang MT, Coyne C, Johnson JT, Stewart AF, Nikiforova MN. Impact of mutational testing on the diagnosis and management of patients with cytologically indeterminate thyroid nodules: a prospective analysis of 1056 FNA samples. J Clin Endocrinol Metab. 2011 Nov;96(11):3390-7. doi: 10.1210/jc.2011-1469. Epub 2011 Aug 31. PMID 21880806
- [Background] Alexander EK, Kennedy GC, Baloch ZW, Cibas ES, Chudova D, Diggans J, Friedman L, Kloos RT, LiVolsi VA, Mandel SJ, Raab SS, Rosai J, Steward DL, Walsh PS, Wilde JI, Zeiger MA, Lanman RB, Haugen BR. Preoperative diagnosis of benign thyroid nodules with indeterminate cytology. N Engl J Med. 2012 Aug 23;367(8):705-15. doi: 10.1056/NEJMoa1203208. Epub 2012 Jun 25. PMID 22731672
- [Background] Ali SZ, Fish SA, Lanman R, Randolph GW, Sosa JA. Use of the afirma(R) gene expression classifier for preoperative identification of benign thyroid nodules with indeterminate fine needle aspiration cytopathology. PLoS Curr. 2013 Feb 11;5:ecurrents.eogt.e557cbb5c7e4f66568ce582a373057e7. doi: 10.1371/currents.eogt.e557cbb5c7e4f66568ce582a373057e7. PMID 23437421
- [Background] Najafzadeh M, Marra CA, Lynd LD, Wiseman SM. Cost-effectiveness of using a molecular diagnostic test to improve preoperative diagnosis of thyroid cancer. Value Health. 2012 Dec;15(8):1005-13. doi: 10.1016/j.jval.2012.06.017. Epub 2012 Sep 25. PMID 23244801
- [Background] Bustin SA, Benes V, Garson JA, Hellemans J, Huggett J, Kubista M, Mueller R, Nolan T, Pfaffl MW, Shipley GL, Vandesompele J, Wittwer CT. The MIQE guidelines: minimum information for publication of quantitative real-time PCR experiments. Clin Chem. 2009 Apr;55(4):611-22. doi: 10.1373/clinchem.2008.112797. Epub 2009 Feb 26. PMID 19246619
- [Background] Pfaffl MW. A new mathematical model for relative quantification in real-time RT-PCR. Nucleic Acids Res. 2001 May 1;29(9):e45. doi: 10.1093/nar/29.9.e45. PMID 11328886
- [Background] Vergara IA, Norambuena T, Ferrada E, Slater AW, Melo F. StAR: a simple tool for the statistical comparison of ROC curves. BMC Bioinformatics. 2008 Jun 5;9:265. doi: 10.1186/1471-2105-9-265. PMID 18534022
- [Background] Melo F, Sali A. Fold assessment for comparative protein structure modeling. Protein Sci. 2007 Nov;16(11):2412-26. doi: 10.1110/ps.072895107. Epub 2007 Sep 28. PMID 17905832
- [Background] Lewis CM, Chang KP, Pitman M, Faquin WC, Randolph GW. Thyroid fine-needle aspiration biopsy: variability in reporting. Thyroid. 2009 Jul;19(7):717-23. doi: 10.1089/thy.2008.0425. PMID 19485775